CLINICAL TRIAL: NCT04278807
Title: Analgesic Efficacy of PENG Block Compared to FIB Block in the Elderly Patient With Fracture of the Proximal Femur in the Emergency Room
Brief Title: PENG-block Versus FIB-block in Emergency Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santo Spirito Hospital, Italy (Other)
Responsible Party: Principal Investigator, Dr Francesco Marrone, Principal Investigator, Santo Spirito Hospital, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSH_PENG_Trial
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Pain Relief in Proximal Femoral Fracture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG-group (Experimental): Ultrasound-guided PENG-block - 30 patients
  Interventions: Procedure: Regional Anesthesia - Nerve Blocks
- FIB-group (Experimental): Ultrasound-guided Fascia Iliaca block - 30 patients
  Interventions: Procedure: Regional Anesthesia - Nerve Blocks

INTERVENTIONS:
Procedure: Regional Anesthesia - Nerve Blocks — Regional Anesthesia and ultrasound-guided nerve blocks

SUMMARY:
The trial aims to verify a possible greater analgesic efficacy of PENG (Pericapsular Nerve Group) block compared to iliac fascia block (FIB block) in elderly patients (age > 65 years) suffering from traumatic fracture of proximal femur in emergency room.

DETAILED DESCRIPTION:
Prospective randomized double-blind single-center preliminary study aimed to demonstrate a possible greater analgesic efficacy of the PENG block compared to the iliac fascia block (FIB block) in elderly patients (age > 65 years) suffering from traumatic fracture of the proximal femur in emergency room.

The study will cover patients aged > 65 years suffering from a proximal traumatic fracture of the femur who access the emergency room of Santo Spirito Hospital in Rome (ASL Roma 1).

ELIGIBILITY:
Inclusion Criteria:

* all patients > 65 years suffering from a proximal traumatic fracture of a femur who access the emergency room of Santo Spirito Hospital in Rome (ASL Rome 1), for whom surgical treatment of osteosynthesis is recommended within 48 hours in accordance with the guidelines of Regional Health System (Regione Lazio).

Exclusion Criteria:

* Failure to acquire written and valid informed consent
* ASA > 3
* Obesity (BMI> 35 kg / m2)
* Contraindications to performing regional anesthesia (severe coagulopathies and / or thrombocytopenia, septic state and / or infections at the block site, allergy to local anesthetics)
* Patients on therapy with antiplatelet agents, anticoagulants or who regularly use opioids, NSAIDs, acetaminophen for chronic painful conditions;
* History of alcohol or drug abuse;
* Severe kidney or liver failure;
* Cognitive alterations, dementia, psychiatric pathologies

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of success rate of PENG block (defined as NRS score </ = 4 at 30 minutes from the blockade placement by comparing it to the analgesic effect of the FIB block, also evaluated at 30 minutes as NRS score </ = 4). | 30 minutes after the placement of nerve block
  Numeric Rating Scale (NRS-score) evaluation, from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Onset time and duration of nerve blockade | from 30 minutes to 12 hours
  First request of analgesic medication after blockade
Evaluation of rest and incident pain | 30 minutes after the placement of nerve block
  Numeric Rating Scale (NRS-score) evaluation, from 0 (no pain) to 10 (worst pain)
Use of rescue-medication in pain treatment | from 30 minutes to 12 hours
  Analgesic drugs administered at the request of the patient in the case of blockade failure
Check for any complications related to analgesic (PENG and FIB) blocks | from 30 minutes to 12 hours
  Recording of any complications related to PENG and FIB blocks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Marrone, Principal Investigator — UOC Anestesia e Rianimazione Santo Spirito Hospital Rome
Locations (1):
- Santo Spirito Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No